CLINICAL TRIAL: NCT05097599
Title: StrataPATH™ (Precision Indications for Approved Therapies): A Study Evaluating the Clinical Activity and Safety of Approved Drugs Within Biomarker-Guided Patients With Solid Tumors
Brief Title: StrataPATH™ (Precision Indications for Approved Therapies)
Acronym: StrataPATH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision and enrollment difficulties
Sponsor: Strata Oncology (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR-004-001; KEYNOTE-F04 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2021-10-01; First posted 2021-10-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Advanced Solid Tumor
Keywords: Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — lorlatinib; encorafenib; binimetinib; talazoparib; sacituzumab govitecan; Axitinib; enfortumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Lorbrena® (lorlatinib) (Other)
  Interventions: Drug: lorlatinib
- Braftovi® (encorafenib) + Mektovi® (binimetinib) (Other)
  Interventions: Drug: encorafenib + binimetinib
- Talzenna® (talazoparib) (Other)
  Interventions: Drug: talazoparib
- Trodelvy® (sacituzumab govitecan-hziy) (Other)
  Interventions: Drug: sacituzumab govitecan
- Inlyta® (axitinib) (Other)
  Interventions: Drug: axitinib
- Enhertu® (fam-trastuzumab deruxtecan-nxki) (Other)
  Interventions: Drug: Fam-Trastuzumab Deruxtecan-Nxki
- Padcev® (enfortumab vedotin) (Other)
  Interventions: Drug: enfortumab vedotin

INTERVENTIONS:
Drug: lorlatinib — This arm of the Strata PATH trial will assess the clinical benefit of Lorbrena® (lorlatinib) in ALK and ROS1 gene fusion positive solid tumors, as detected by Strata testing, with the exception of NSCLC.
  Arms: Lorbrena® (lorlatinib)
Drug: encorafenib + binimetinib — This arm of the Strata PATH trial will assess the clinical benefit of Braftovi® (encorafenib) + Mektovi® (binimetinib) in BRAF p.v600X mutated solid tumors, as detected by Strata testing, with the exception of melanoma and colorectal cancer.
  Arms: Braftovi® (encorafenib) + Mektovi® (binimetinib)
Drug: talazoparib — This arm of the Strata PATH trial will assess the clinical benefit of Talzenna® (talazoparib) in patients with advanced solid tumors harboring deep deletions or deleterious mutations with LOH in BRCA1/2 and PALB2, as detected by Strata testing, excluding HER2 negative breast cancer.
  Arms: Talzenna® (talazoparib)
Drug: sacituzumab govitecan — This arm of the Strata PATH trial will assess the clinical benefit of Trodelvy® (sacituzumab govitecan) in patients with advanced solid tumors and are Trop2 Treatment Response Score High (Trop2 TRS-H), as detected by Strata testing, excluding triple negative breast cancer, hormone receptor positive/ human epidermal growth factor receptor 2 negative (HR+/HER2-) breast cancer, metastatic urothelial cancer, non-small cell lung (NSCLC) cancer, small cell lung cancer (SCLC), head and neck cancer, colorectal cancer (CRC), and endometrial cancer.
  Arms: Trodelvy® (sacituzumab govitecan-hziy)
Drug: axitinib — This arm of the Strata PATH trial will assess the clinical benefit of Inlyta® (axitinib) in patients with advanced solid tumors and are Angiogensis Inhibitor Treatment Response Score High (Angio TRS-H), as detected by Strata testing, excluding renal cell carcinoma, alveolar soft part sarcoma, and solitary fibrous tumors.
  Arms: Inlyta® (axitinib)
Drug: Fam-Trastuzumab Deruxtecan-Nxki — This arm of the Strata PATH trial will assess the clinical benefit of Enhertu ® in patients with advanced solid tumors with Her2 overexpression
  Other Names: Enhertu
  Arms: Enhertu® (fam-trastuzumab deruxtecan-nxki)
Drug: enfortumab vedotin — This arm of the Strata PATH trial will assess the clinical benefit of Padcev® in patients with advanced solid tumors with nectin-4 overexpression
  Other Names: Padcev
  Arms: Padcev® (enfortumab vedotin)

SUMMARY:
StrataPATH™ is a non-randomized, open-label trial designed to explore efficacy and safety of multiple FDA-approved and commercially available cancer therapies in new, biomarker-guided patient populations.

DETAILED DESCRIPTION:
StrataPATH is a non-randomized, open-label trial designed to explore efficacy and safety of multiple FDA-approved and commercially available cancer therapies in new, biomarker-guided patient populations. Aiming to increase clinical benefit for patients, this study will leverage technology advancements, scientific literature, and Strata's real-world evidence to define novel, highly responsive pan-tumor molecular indications for FDA-approved therapies in both the advanced and micro-metastatic settings. Strata will rapidly identify participants who have efficacy signals for possible expansion into adaptive or randomized studies. Enrollment in each drug/biomarker cohort is competitive. Cohorts may be added, changed, or discontinued over the course of the study

ELIGIBILITY:
To be eligible to participate in this study, an individual must meet each of the criterion below and the criteria indicated in the selected biomarker/drug cohort appendix:

1. Male or female ≥18 years of age.
2. Pathologically confirmed solid tumor
3. Participants must be able to follow study visit schedule and willing to provide up to 20 mL of peripheral blood samples at the indicated time points
4. CGP results need to be from a test conducted in a CLIA approved laboratory and archival formalin-fixed, paraffin-embedded (FFPE) tumor tissue is required for confirmatory testing of non-Strata test results unless otherwise indicated within the cohort-specific protocol criteria.
5. Biomarker positive for the defined cohort
6. For individuals with non-primary, treated or stable brain metastases: No evidence of progression (defined as no radiographic evidence of progression) for at least 4 weeks prior to consent.
7. Adequate bone marrow, organ function & laboratory parameters as determined by the treating physician unless otherwise indicated within the cohort-specific protocol criteria.
8. Adequate cardiac function: 1) Left ventricular ejection fraction (LVEF) ≥ 50% and 2) QTc interval ≤ 470 ms (females) or ≤ 450 ms (males) average preferred.

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Receiving another cancer treatment
2. Major surgery within 4 weeks prior to study entry
3. Has received a systemic cancer treatment within 3 weeks of first study dose
4. Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers that have been diagnosed and treated within the past 3 years are eligible: cervical/prostate carcinoma in situ, superficial bladder cancer, non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 3 years and felt to be at low risk of recurrence should be discussed with the study principal investigator to determine eligibility.
5. Participant has primary central nervous system tumor.
6. A woman of childbearing potential who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Females who are pregnant or nursing or plan to become pregnant or anyone unwilling to use contraception for the duration of treatment.
8. Ongoing toxicity of CTCAE grade >2, other than peripheral neuropathy, related to anticancer therapy that was completed within 4 weeks of consent.
9. Ongoing peripheral neuropathy of CTCAE grade >3.
10. History of stroke including transient ischemic attack (TIA) or acute myocardial infarction within 6 months of consent.
11. Participant has a known history of human immunodeficiency virus (HIV), Hepatitis B or known active Hepatitis C virus infection.
12. Medical condition that would place the patient at risk as a result of blood donation, such as bleeding disorder.
13. Any other clinically significant medical condition that, in the opinion of the treating physician, makes participation undesirable, including but not limited to ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) defined as the percentage of participants with a best overall response of CR or PR based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as assessed by the investigator | Assessed throughout end of study, up to 5 years
  RECIST criteria will be used to assess the clinical activity of cancer treatments in participants with pre-specified biomarker profiles.

SECONDARY OUTCOMES:
Duration of Response (DoR) defined as the time from first documentation of disease response (CR or PR) until first documentation of progressive disease | Assessed throughout end of study, up to 5 years
  DoR will be used to assess the duration of response of cancer treatments in participants with pre-specified biomarker profiles.
Time to Treatment Discontinuation (TTD) defined as length of time from the date the participant initiates the systemic treatment to the date the participant discontinues treatment as compared to prior TTD from prior cancer treatment | Assessed throughout end of study, up to 5 years
  TTD will be used to assess the duration of response of cancer treatments in participants with pre-specified biomarker profiles.
TTnT (Time to Next Treatment) defined as the length of time from the date the participant initiates study treatment to the date the participant initiates their next systemic treatment or death. | Assessed throughout end of study, up to 5 years
  TTnT will be used to assess the duration of response of cancer treatments in participants with pre-specified biomarker profiles.
ctDNA response: The proportion of participants with a <50% ratio of mean variant allele frequency (VAF) will be defined as ctDNA responders | 6 months
  Molecular response calculated as a ratio of mean VAF on treatment at 6 months compared to baseline VAF will be used to assess the clinical activity of cancer treatments in participants with pre-specified biomarker profiles.
Overall Survival (OS) | Assessed throughout end of study, up to 5 years
  Evaluate overall survival (OS) for participants who received a cancer treatment with pre-specified biomarker profiles
Incidence of serious adverse events (SAEs) | Assessed throughout end of study, up to 5 years
  Monitor and summarize any unexpected safety events in participants who received a biomarker-guided cancer treatment
ctDNA Response Rate | Assessed throughout end of study, up to 5 years
  Evaluate ctDNA response rate at additional timepoints for participants who received cancer treatment with pre-specified biomarker profiles

OTHER OUTCOMES:
Explore the correlation between serial ctDNA levels over time and participant response to cancer therapy based on RECIST 1.1, as assessed by the investigator. | Assessed throughout end of study, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kat Kwiatkowski, PhD, Study Director — Strata Oncology
Locations (4):
- United States (4):
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Kettering Health Network, Kettering, Ohio
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Ramalingam SS, Yang JC, Lee CK, Kurata T, Kim DW, John T, Nogami N, Ohe Y, Mann H, Rukazenkov Y, Ghiorghiu S, Stetson D, Markovets A, Barrett JC, Thress KS, Janne PA. Osimertinib As First-Line Treatment of EGFR Mutation-Positive Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Mar 20;36(9):841-849. doi: 10.1200/JCO.2017.74.7576. Epub 2017 Aug 25. PMID 28841389
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Khozin S, Miksad RA, Adami J, Boyd M, Brown NR, Gossai A, Kaganman I, Kuk D, Rockland JM, Pazdur R, Torres AZ, Zhi J, Abernethy AP. Real-world progression, treatment, and survival outcomes during rapid adoption of immunotherapy for advanced non-small cell lung cancer. Cancer. 2019 Nov 15;125(22):4019-4032. doi: 10.1002/cncr.32383. Epub 2019 Aug 5. PMID 31381142
- [Background] Blumenthal GM, Gong Y, Kehl K, Mishra-Kalyani P, Goldberg KB, Khozin S, Kluetz PG, Oxnard GR, Pazdur R. Analysis of time-to-treatment discontinuation of targeted therapy, immunotherapy, and chemotherapy in clinical trials of patients with non-small-cell lung cancer. Ann Oncol. 2019 May 1;30(5):830-838. doi: 10.1093/annonc/mdz060. PMID 30796424
- [Background] Prentice RL. Surrogate endpoints in clinical trials: definition and operational criteria. Stat Med. 1989 Apr;8(4):431-40. doi: 10.1002/sim.4780080407. PMID 2727467
- [Background] Fleming TR, Powers JH. Biomarkers and surrogate endpoints in clinical trials. Stat Med. 2012 Nov 10;31(25):2973-84. doi: 10.1002/sim.5403. Epub 2012 Jun 18. PMID 22711298
- [Background] Thompson JC, Carpenter EL, Silva BA, Rosenstein J, Chien AL, Quinn K, Espenschied CR, Mak A, Kiedrowski LA, Lefterova M, Nagy RJ, Katz SI, Yee SS, Black TA, Singh AP, Ciunci CA, Bauml JM, Cohen RB, Langer CJ, Aggarwal C. Serial Monitoring of Circulating Tumor DNA by Next-Generation Gene Sequencing as a Biomarker of Response and Survival in Patients With Advanced NSCLC Receiving Pembrolizumab-Based Therapy. JCO Precis Oncol. 2021 Mar 19;5:PO.20.00321. doi: 10.1200/PO.20.00321. eCollection 2021. PMID 34095713
- [Background] Zhang Q, Luo J, Wu S, Si H, Gao C, Xu W, Abdullah SE, Higgs BW, Dennis PA, van der Heijden MS, Segal NH, Chaft JE, Hembrough T, Barrett JC, Hellmann MD. Prognostic and Predictive Impact of Circulating Tumor DNA in Patients with Advanced Cancers Treated with Immune Checkpoint Blockade. Cancer Discov. 2020 Dec;10(12):1842-1853. doi: 10.1158/2159-8290.CD-20-0047. Epub 2020 Aug 14. PMID 32816849
- [Background] Jung SH, Lee T, Kim K, George SL. Admissible two-stage designs for phase II cancer clinical trials. Stat Med. 2004 Feb 28;23(4):561-9. doi: 10.1002/sim.1600. PMID 14755389
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- See also: American Cancer Society Cancer Statistics Center, 2020 9/4/2020 — https://cancerstatisticscenter.cancer.org/#/.
- See also: U.S. Food and Drug Administration, FDA grants accelerated approval to pembrolizumab for first tissue/site agnostic indication. 2017. — https://www.fda.gov/drugs/resources-information-approved-drugs/fda-grants-accelerated-approval-pembrolizumab-first-tissuesite-agnostic-indication
- See also: Merck, Merck's KEYTRUDA® (pembrolizumab) Demonstrated Superior Disease-Free Survival (DFS) Compared With Placebo as Adjuvant Therapy in Patients With Renal Cell Carcinoma (RCC) Following Surgery, in Press Release. 2021. — https://www.merck.com/news/mercks-keytruda-pembrolizumab-demonstrated-superior-disease-free-survival-dfs-compared-with-placebo-as-adjuvant-therapy-in-patients-with-renal-cell-carcinoma-rcc-following-surgery/
- See also: Temple, R., A regualtory authority's opinion about surrogate endpoints, in Clinical Measurement in Drug Evaluation, W.T. Nimmo, Editor. 1995, J.Wiley: New York. — http://scholar.google.com/scholar_lookup?&title=Clinical%20Measurement%20in%20Drug%20Evaluation&pages=3-22&publication_year=1995&author=Temple%2CRJ
- See also: U.S. Food and Drug Administration, Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics Guidance for Industry. 2018. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/clinical-trial-endpoints-approval-cancer-drugs-and-biologics
- See also: U.S. Food and Drug Administration, FDA approves larotrectinib for solid tumors with NTRK gene fusions. 2018. — https://www.fda.gov/drugs/fda-approves-larotrectinib-solid-tumors-ntrk-gene-fusions

DOCUMENTS (1):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT05097599/Prot_000.pdf